CLINICAL TRIAL: NCT01068977
Title: A Phase I, Open Label, Dose Escalation Study of the Safety and Pharmacology of MetMAb (PRO143966), a Monovalent Antagonist Antibody to the Receptor C-Met, Administered Intravenously in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of the Safety and Pharmacology of MetMAb (PRO143966), a Monovalent Antagonist Antibody to the Receptor C-Met, Administered Intravenously in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OAM4224g
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Solid Cancers
MeSH Terms: interventions — Bevacizumab; onartuzumab

ARMS (3):
- Stage I (Experimental)
  Interventions: Drug: MetMAb
- Stage II (Experimental)
  Interventions: Drug: MetMAb
- Stage III (Experimental)
  Interventions: Drug: bevacizumab; Drug: MetMAb

INTERVENTIONS:
Drug: bevacizumab — Repeating intravenous dose
  Arms: Stage III
Drug: MetMAb — Repeating escalating intravenous dose
  Arms: Stage I; Stage III
Drug: MetMAb — Repeating intravenous dose
  Arms: Stage II

SUMMARY:
This is a Phase I, open label, dose-escalation study of MetMAb administered by intravenous (IV) infusion in patients with advanced solid malignancies that are refractory to or for which there is no standard of care. The study consists of a dose-escalation stage, an expansion stage testing MetMAb at the recommended Phase II dose (RP2D), and a dose-escalation stage testing the combination of MetMAb, at two different doses with bevacizumab at a recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of incurable, locally advanced, or metastatic solid malignancy that has failed to respond to at least one prior regimen or for which there is no standard therapy
* Disease that is measurable or evaluable by Response Evaluation Criteria In Solid Tumors (RECIST)
* Life expectancy ≥12 weeks

Exclusion Criteria:

* Less than 4 weeks since the last anti-tumor therapy
* Patients receiving erythropoietin products
* Active infection requiring antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs
* Symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Clinically important history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus infection
* Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MetMAb alone or in combination with bevacizumab will be assessed (frequency and nature of dose-limiting toxicities; nature, severity, and relatedness of adverse events; changes in vital signs and clinical laboratory parameters) | Length of study

SECONDARY OUTCOMES:
Objective response, defined as a complete or partial response confirmed ≥4 weeks after initial documentation | Length of study
Duration of objective response | Length of study
Progression-free survival | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Premal Patel, M.D., Study Director — Genentech, Inc.